CLINICAL TRIAL: NCT02420067
Title: An International Collaborative Study: Screening for Endolymphatic Sac Tumours (ELSTs) in Von Hippel-Lindau (vHL) Patients
Brief Title: Screening for Endolymphatic Sac Tumours (ELSTs) in Von Hippel-Lindau (vHL) Patients
Status: Recruiting | Type: Observational
Sponsor: Marie Luise Bisgaard, MD (Other)
Collaborators: Rigshospitalet, Denmark (Other); St Thomas' Hospital, London (Other); Fundación Hospital de Madrid (Other); National Cancer Centre, Singapore (Other); Yokosuka City Shimin Hospital (Other); Amrita Institute of Medical Sciences & Research Center (Other)
Responsible Party: Sponsor-Investigator, Marie Luise Bisgaard, MD, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: H-A-2007-0125, A
Record Dates: First submitted 2015-04-09; First posted 2015-04-17 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Von Hippel-Lindau Disease
Keywords: von Hippel-Lindau disease; Endolymphatic sac tumors; Audiological examination; MRI; Surveillance
MeSH Terms: conditions — von Hippel-Lindau Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to investigate how best to screen for Endolymphatic sac tumors (ELSTs) in von Hippel-Lindau (vHL) patients in order to diagnose the ELSTs while they are still small so that hearing loss can be prevented.

Up to 16% of vHL patients are known to develop endolymphatic sac tumors in the inner ear that can cause permanent hearing loss. However, the ELSTs are often not found before hearing loss has already occurred. The challenge for doctors is to diagnose the ELSTs at early stages before they cause often irreversible deafness. In order to find ELSTs before they cause hearing loss, it is important to screen for the tumors prophylactically, that is screen all vHL patients regardless of whether or not they have symptoms.

Who can join? Persons diagnosed with vHL who are at least 15 years old. The investigators include patients WITH OR WITHOUT a diagnosed ELST.

What does it involve? You need to have a hearing test and an MRI of the brain, where the inner ear can be seen, most vHL patients have already had this done as part of their surveillance program.

Participants will be asked to participate in follow up examinations (hearing test and/or MRI of the brain) after 2, 5, and 10 years.

How can I join? A doctor has to be responsible for the study in each country where vHL patients participates.

Ask the doctor who manages your vHL examinations to contact us or contact us yourself and the investigators will help you find a doctor in your country who will participate in the study.

DETAILED DESCRIPTION:
Background:

von Hippel-Lindau disease (vHL) is a hereditary multi-system disease requiring life-long prophylactic surveillance. Affected individuals are predisposed to development of tumors and cysts in multiple organs. In recent years, it has become apparent that endolymphatic sac tumors (ELSTs), aggressive tumors of the petrous bone, occur in up to 16% of vHL patients. ELST can lead to severe and progressive hearing loss and vertigo as well as other audio-vestibular and neurological symptoms. However, surgical excision of tumors can preserve patients' pre-operative hearing level, and eliminate most other audio-vestibular symptoms. As even small ELSTs have been shown to lead to sudden and irreversible deafness, timely diagnosis of ELSTs is essential to prevent severe audio-vestibular morbidity in ELST patients. Several recommendations of ELST surveillance in vHL patients have been proposed; some suggest that diagnostic tests for ELST should be done only in vHL patients with subjective audio-vestibular symptoms, while others recommend audiological examinations or MRI of the inner ear in all vHL patients as a screening tool. However, there has not previously been much focus on specification of screening strategies, and it is not known, which is the most optimal approach. The results of a national study of ELST surveillance among Danish vHL patients indicated that specific patterns of audiologic parameters in patients with ELSTs, indicating that a distinct audiologic pattern may be typical in ELST development, perhaps even before the ELST is detectable on MRI. However, a larger study of audiologic parameters in vHL patients with and without diagnosed ELSTs is needed in order to fully investigate such a model and its use in early ELST detection.

Objective The overall objective of this study is to establish audiologic characteristics among vHL patients with and without ELST, and investigate whether specific patterns in audiometric parameters correspond to different stages in ELST development.

Material and Methods:

The study is a multi-center prospective cohort study that includes adult vHL patients, who are followed with clinical interviews about subjective audio-vestibular symptoms, MRI of the inner ear, and audiometry.

Results of all subjects' audiological and radiologic examinations will be collected at the Department of Cellular and Molecular Medicine, University of Copenhagen. Results will be blinded with regard to ELST history and radiologic results and evaluated by a single senior ear-nose-and-throat specialist, who will look for specific patterns in audiologic parameters over time. Radiologic images will be blinded with regard to symptoms and audiological examination results and will be evaluated by a single radiology specialist, who will look only at the inner ear and surrounding structures for presence of imaging-visible ELSTs and evaluate size and pattern of growth of ELSTs if possible. Audiometric characteristics will be correlated with presence of MRI visible ELSTs and patients' subjectively reported audio-vestibular symptoms to determine whether specific patterns of audiological parameters are distinct for ELSTs and their stages of tumor growth.

A followed-up of all study participants is planned after 2, 5 and 10 years after patients' last assessed audiological examinations included in the initial study.

The initiators of the project are responsible for evaluation and analysis of data, and are required to inform local project managers of any differences in their evaluation of examinations compared to the local evaluations of the same examinations.

Local project managers are required to inform all of their local participants the results of their examinations. If any ELSTs are found in participants, local project managers must offer management of the ELSTs according to local recommendations. The initiators of the project will offer help and counseling in relation to ELST management and treatment if necessary.

Considerations of biomedical research ethics:

The Danish part of the study has been approved by the Danish Regional Committees on Biomedical Research, who have also approved that results from all participating institutions outside of Denmark can be collected and analyzed in Denmark. Each participating institution outside of Denmark must make sure that the study is also approved according to regional law. Oral and written consent must be obtained from all subjects, and results must be coded before data is sent to Denmark for analysis.

Data management:

The investigators have approval for the study from the Danish Data Protection Agency. All data analysis will take place under the University of Copenhagen in Denmark.

Significance and perspectives:

The present study will clarify the significance of audiologic examination in ELST surveillance and improve ELST screening for vHL patients.

Publication:

The results will be published in international, scientific journals. Collaborators will be included ad co-authors in any publications of the results of this study according to Vancouver rules.

Funding:

The project is financially supported as a subproject of a larger PhD project. Salary of the PhD student, Marie Louise Mølgaard Binderup is financed by the Danish Cancer Society with approximately181,000 Euros, while the expenses of operation of the PhD project is supported by the Lundbeck Foundation with approximately 65,000 Euros, of which approximately 4,000 Euros is estimated to be used for expenses of the present subproject. The supporting organisations solely provide financial support and have no influence on study design, the execution of study, or publication of results. Initiators of this project will not apply for further financial support for this subproject.

Collaborating institutions and participating patients will not receive any financial support from the mentioned sources.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of vHL (either a carrier of a VHL mutation or vHL diagnosed by clinical criteria, i.e. at least two vHL-related manifestations diagnosed or one vHL-related manifestation diagnosed AND a first-degree relative with vHL)
* At least one audiological examination (including an audiogramme) and one MRI examination of the brain also visualizing the inner ear within 12 months of each other

Exclusion Criteria:

* Children under the age of 15 years

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: vHL patients, with or without a diagnosed ELST, who have had at least one audiological examination AND one MRI of the brain and inner ear within a 12 month period
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2011-02; Primary Completion 2017-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
In each ear: development of an ELST during the study period correlated to baseline hearing level. | Change in status of ELST diagnosis from during the ten year period from study baseline to study end.
  Presence and size of an ELST as diagnosed by an MRI at any time during the study period correlated to the baseline hearing level in the ear as defined by hearing level in decibel in air- and bone conduction at predefined frequencies 125, 250, 500, 1000, 2000, 4000, 8000 Hz measured with pure-tone audiometry.

SECONDARY OUTCOMES:
In each ear: development of an ELST during the study period correlated to hearing level at two year follow-up. | Change in status of ELST diagnosis from during the 8 year period from two year follow-up to study end.
  Presence and size of an ELST as diagnosed by an MRI at any time during the study period correlated to the hearing level at the two year follow-up in the ear as defined by hearing level in decibel in air- and bone conduction at predefined frequencies 125, 250, 500, 1000, 2000, 4000, 8000 Hz measured with pure-tone audiometry.
In each ear: development of an ELST during the study period correlated to hearing level at five year follow-up. | Change in status of ELST diagnosis from during the 5 year period from five year follow-up to study end.
  Presence and size of an ELST as diagnosed by an MRI at any time during the study period correlated to the hearing level at the five year follow-up in the ear as defined by hearing level in decibel in air- and bone conduction at predefined frequencies 125, 250, 500, 1000, 2000, 4000, 8000 Hz measured with pure-tone audiometry.
In each ear: development of an ELST during the study period correlated to presence of low-frequency hearing loss (sensorineural) pattern A at baseline assessment. | Change in status of ELST diagnosis during the 10 year period from study initiation to study end.
  Presence and size of an ELST as diagnosed by an MRI at any time during the study period correlated to presence of low-frequency hearing loss (sensorineural) type A as defined by (Th500 Hz - Th1.000 Hz > 5 dB) AND (Th250 Hz > Th1.000 Hz) measured during a pure-tone audiometry at baseline assessment.
In each ear: development of an ELST during the study period correlated to presence of low-frequency hearing loss (sensorineural) pattern A at the two-year follow-up assessment.. | Change in status of ELST diagnosis during the 8 year period from study initiation to the two-year follow-up assessment.
  Presence and size of an ELST as diagnosed by an MRI at any time during the study period correlated to presence of low-frequency hearing loss (sensorineural) type A as defined by (Th500 Hz - Th1.000 Hz > 5 dB) AND (Th250 Hz > Th1.000 Hz) measured during a pure-tone audiometry at two-year follow-up assessment.
In each ear: development of an ELST during the study period correlated to presence of low-frequency hearing loss (sensorineural) pattern A at the five-year follow-up assessment. | Change in status of ELST diagnosis during the 5 year period from study initiation to the five-year follow-up assessment.
  Presence and size of an ELST as diagnosed by an MRI at any time during the study period correlated to presence of low-frequency hearing loss (sensorineural) type A as defined by (Th500 Hz - Th1.000 Hz > 5 dB) AND (Th250 Hz > Th1.000 Hz) measured during a pure-tone audiometry at five-year follow-up assessment.
In each ear: development of an ELST during the study period correlated to presence of low-frequency hearing loss (sensorineural) pattern B at baseline assessment. | Change in status of ELST diagnosis during the 10 year period from study initiation to study end.
  Presence and size of an ELST as diagnosed by an MRI at any time during the study period correlated to presence of low-frequency hearing loss (sensorineural) type B as defined by (Th1.000 Hz > Th2.000 Hz) and (Th500 - Th2.000 Hz > 9 dB) and (Th250 Hz -2.000 H< > 9 dB) measured during a pure-tone audiometry at baseline assessment.
In each ear: development of an ELST during the study period correlated to presence of low-frequency hearing loss (sensorineural) pattern B at the two-year follow-up assessment. | Change in status of ELST diagnosis during the 8 year period from study initiation to the two-year follow-up assessment.
  Presence and size of an ELST as diagnosed by an MRI at any time during the study period correlated to presence of low-frequency hearing loss (sensorineural) type B as defined by (Th1.000 Hz > Th2.000 Hz) and (Th500 - Th2.000 Hz > 9 dB) and (Th250 Hz -2.000 H< > 9 dB) measured during a pure-tone audiometry at the two-year follow-up assessment.
In each ear: development of an ELST during the study period correlated to presence of low-frequency hearing loss (sensorineural) pattern B at the five-year follow-up assessment. | Change in status of ELST diagnosis during the 5 year period from study initiation to the five-year follow-up assessment.
  Presence and size of an ELST as diagnosed by an MRI at any time during the study period correlated to presence of low-frequency hearing loss (sensorineural) type B as defined by (Th1.000 Hz > Th2.000 Hz) and (Th500 - Th2.000 Hz > 9 dB) and (Th250 Hz -2.000 H< > 9 dB) measured during a pure-tone audiometry at the five-year follow-up assessment.
Development of an ELST during the study period correlated to presence of subjective audio-vestibular symptoms at the baseline assessment. | Change in status of ELST diagnosis during the 10 year period from study initiation to the study end.
  Presence and size of an ELST as diagnosed by an MRI at any time during the study period correlated to presence of audio-vestibular symptoms in the form of hearing loss, tinnitus, vertigo, sense of aural fullness, and ear pain that are not known to have an non-ELST cause as reported by the patient at the baseline assessment.
Development of an ELST during the study period correlated to presence of subjective audio-vestibular symptoms at the two-year follow-up assessment. | Change in status of ELST diagnosis during the 8 year period from study initiation to the two-year follow-up assessment.
  Presence and size of an ELST as diagnosed by an MRI at any time during the study period correlated to presence of audio-vestibular symptoms in the form of hearing loss, tinnitus, vertigo, sense of aural fullness, and ear pain that are not known to have an non-ELST cause as reported by the patient at the two-year follow-up assessment.
Development of an ELST during the study period correlated to presence of subjective audio-vestibular symptoms at the five-year follow-up assessment. | Change in status of ELST diagnosis during the 5 year period from study initiation to the five-year follow-up assessment.
  Presence and size of an ELST as diagnosed by an MRI at any time during the study period correlated to presence of audio-vestibular symptoms in the form of hearing loss, tinnitus, vertigo, sense of aural fullness, and ear pain that are not known to have an non-ELST cause as reported by the patient at the five-year follow-up assessment.

OTHER OUTCOMES:
VHL mutation status related to presence of hearing loss and/or presence of ELST at any time during the study. | Assessed at the end of the study ten year after study initiation.
  Presence of a VHL mutation confirmed by molecular analysis correlated to hearing loss as determined during audiometry and/or to presence of an ELST as diagnosed by MRI during the study.
Type of VHL mutation related to presence of hearing loss and/or presence of ELST at any time during the study. | Assessed at the end of the study ten year after study initiation
  Type of a VHL mutation confirmed by molecular analysis (mutations predicted to truncate the protein product or not) correlated to hearing loss as determined during audiometry and/or to presence of an ELST as diagnosed by MRI during the study.
Type of clinical vHL type related to presence of hearing loss and/or presence of ELST at any time during the study. | Assessed at the end of the study ten year after study initiation
  Type of clinical vHL type as defined by previously diagnosis of other types of vHL-related manifestations in the patient (cerebellar hemangioblastomas, retinal hemangioblastoma, renal cell carcinoma, renal cysts, pancreatic tumors, pancreatic cysts, pheochromocytomas, paragangliomas, Epidydydimal cysts/ cysts of the broad uterine ligament) correlated to hearing loss as determined during audiometry and/or to presence of an ELST as diagnosed by MRI during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Luise Bisgaard, M.D., Principal Investigator — Department of Cellular and Molecular Medicin, University of Copenhagen
Locations (1):
- Department of Cellular and Molecular Medicine, University of Copenhagen, Copenhagen, Copenhagen N, Denmark